CLINICAL TRIAL: NCT01589640
Title: Phase 4 Study Accessing Patient Satisfaction and Tear Osmolarity While Using Blink Tears, Blink Gel Tears and Systane Balance
Brief Title: Patient Satisfaction and Tear Osmolarity With the Use of Blink Tears, Blink Gel Tears and Systane Balance
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ophthalmic Consultants of Connecticut (Other)
Responsible Party: Sponsor
Other Study IDs: EDD-BLNK-12-001
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Polyethylene Glycols; Propylene Glycol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Blink Tears: Blink Tears is an over the counter artificial tear
  Interventions: Other: Blink Tears lubricating Eye Drops
- Blink Gel Tears: Blink Gel Tears is an over the counter artifical tear product
  Interventions: Other: Blink Gel Tears Lubricating Eye Drops
- Systane Balance: Systane Balance is an over the counter artificial Tear product
  Interventions: Other: Systane Balance Lubricant Eye Drop

INTERVENTIONS:
Other: Blink Tears lubricating Eye Drops — 2 drops per eye drosed four times per day (8:00 Am, 12:00 PM, 4:00 PM and 8:00 PM)
  Other Names: Blink Tears
  Groups: Blink Tears
Other: Blink Gel Tears Lubricating Eye Drops — 2 drops per eye dosed four times per day (8:00 AM, 12:00PM, 4:00 PM and 8:00 PM)
  Other Names: Blink Gel Tears
  Groups: Blink Gel Tears
Other: Systane Balance Lubricant Eye Drop — 2 Drops per eye dosed four times per day ( 8:00 AM, 12:00 PM, 4:00 PM and 8:00PM)
  Other Names: Systane Balance
  Groups: Systane Balance

SUMMARY:
This is a single center clinical study designed to determine patient satisfaction and the effect of the use of artificial tears on tear osmolarity with time after instillation of three commercially available artifical tear eye solutions ( Blink Tears, Blink Gel Tears and Systane Balance).

DETAILED DESCRIPTION:
Patient satisfaction and tear osmolarity with the use of Blink Tears, Blink Gel Tears and Systane Balance.

ELIGIBILITY:
Inclusion Criteria:

* male or femal subjects (aged 18 or older)
* diagnosed with mild to moderate dry eye syndrome
* provide written informed consent and sign/date a health information release
* women of childbreaing potential must be willing to practice effective contraception for the duration of the study.

Exclusion Criteria:

* have any active ocular disease other than mild to moderate dry eye sundrome that would interfere with study interpretation
* active ocular allergy in any eye
* history of or active ocular infection/inflammation
* concomitant use of contact lenses (unilateral or bilateral)
* history of any corneal refractive laser surgery (e.g., LASIK, LASEK, RK,PRK) in the study eye (s);
* corneal disorder or abnormality that affects cornea sensitivity or normal spreading of the tear film in any eye.
* history of any intaocular surgery or glaucoma laser surgery (e.g., ALT, SLT) in the study eye (s)
* known sensitivity or allergy to any of the study medications or their components;
* uncontrolled systemic disease;
* contraindication to pupil dilation;
* Schirmer's Test- Standard Test (with anesthesia) result of less than or equal to 3 MM
* use of artifical tears prior to Baseline Visit (Visit 2, Day 0);
* Current use, use within 2 weeks prior to Baseline Visit ( Visit 2,Day 0) or likely use during the study period of any topical ophthalmic medications (e.g., antibotics, glaucoma medications) other than ophthalmic medications used in the study.
* use of any omega 3 supplement, artificial tear product (s), vasoconstrictor and/or redness reliever ocular drops 30 days prior to or during the study perior;
* use of cyclosporine ocular drops 12 months prior to or will require ocular surgery during the study period.
* females who are pregnany, nursing or planning a pregnancy or who are of childbearing potenital and not using a reliable method of contraception;
* any systemic disease or clinical evidence of any condition which would make the subject, in the opinion of the investigator, unsuitable for the study or could potentially confound the study results; and
* concurrent participation or prior participation in any investigational drug or device study within the last 30 days prior to the Screening Visit (Visit 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: greater then age 18
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy variable is tear osmolarity | 28 days

SECONDARY OUTCOMES:
Secondary efficacy variable is the Patient Symptom Questionnaire | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Eric Donnenfeld, M.D., Principal Investigator — Ophthalmic Consultants of Connecticut
Locations (1):
- Ophthalmic Consultants of Connecticut, Fairfield, Connecticut, United States